CLINICAL TRIAL: NCT02894346
Title: Moving Towards Learning: Understanding Teachers' Motivation for Using Physical Activity as a Tool for Learning
Brief Title: Moving Towards Learning: Understanding Teachers' Motivation
Acronym: MTL
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Louise Stjerne Knudsen, Ph.d. student, University of Southern Denmark
Other Study IDs: SDUSF-2015-147/R1
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Motivation
Keywords: Motivation; Teachers; Physical activity; School
MeSH Terms: conditions — Motor Activity | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Teachers: Public school teachers in Denmark - across age, gender, subject, class and experience.
  Interventions: Other: Teachers

INTERVENTIONS:
Other: Teachers — Teachers are exposed to the WTMST survey that based on the theory of Self-Determination (SDT) will categorize them according to the elements of the SDT: Intrinsic, identified, introjected, external and a motivation.
  Other Names: The Work Task Motivation Scale for Teachers (WTMST)

SUMMARY:
Since 2014 45 minutes of physical activity (PA) has been a mandatory part of all public schools in Denmark. PA has to be part of subject teaching, including Physical Education (PE), and of so-called support teaching. Research has shown that teachers not always find it meaningful to implement PA during lessons. In addition, even though PA seemingly has positive impacts on children's concentration and learning, teachers find it hard to integrate good quality PA with the learning objectives of any school subject. The purpose of this study is therefore to: 1) Analyse teachers' underlying factors of motivation for using PA as a learning tool using The Self Determination Theory (SDT), and 2) analyse how to support teachers' motivation by using the theory of scaffolding.

The study uses mixed methods. Through quantitative and qualitative methods the study analyses behavioural patterns focusing on teachers' motivation for implementing PA and need for support. The process is iterative moving from a quantitative (survey) to a qualitative approach (interviews).

The study provides new and important knowledge of teachers' motivation for implementing PA as a learning tool. Results from SDT analysis will point out teachers' levels of controlled versus autonomous motivation, and analysing teacher's need for scaffolding will give insight into how teachers' motivation can be framed in the process of implementing PA.

There can be both potentials and barriers for implementing PA in a learning context, and in the process of implementing PA during school days the role of the teacher becomes crucial. It is therefore important to understand teachers underlying factors of motivation for using PA as a learning tool, and in order to help them carry out qualified and suitable PA, it is important that the investigators know how to support them and maintain their motivation in this process.

DETAILED DESCRIPTION:
Introduction According to research there is a positive link between physical activity and academic performance in children and young people, which means that exercise not only benefit physical health and well-being, but also cognition and performance in a learning context. However, developing and engaging in physical activity (PA) requires motivation and most importantly research shows that people who are intrinsically motivated are more likely to engage in PA consistently. When integrating PA in a school context the role of the teacher becomes crucial, as the teacher is responsible for developing and carrying out qualified PA activities. It is therefore important to understand the underlying factors of motivation - especially teachers' motivation for using PA as a tool for learning.

There can be both potential and barriers for integrating PA in a learning context. A recent study from the University of Southern Denmark suggests that teachers are willing to implement PA, and that it can be, but not always is, meaningful to use in a school setting and as a tool for learning. Furthermore, a number of teachers believe that PA and PE activities have a positive impact on concentration and learning, however, they find it hard to integrate and carry out qualified PA activities with suitable learning objectives during school lessons. The study also suggests that implementing PA as a tool for learning depends on how much teachers know about the didactics in relation to using PA.

With the implementation of The Danish School Reform in 2014, PA became a mandatory part of the school day, stating that all children must engage in at least 45 minutes of daily activity. The 45 minutes must either be part of the pupils learning process or separately from subject and lessons. It is, however, not stated in the reform what kind of activity, of what intensity, and at what time during the school day PA must be carried out. The reform is therefore open to interpretation and can be perceived by teachers in many ways. As a consequence schools and teachers carry out the 45 minutes of daily activity very differently - not only based on the lack of information in the Reform, but also based on their experience with and knowledge of PA. It is therefore important to examine and understand how teachers can be supported in the process of using PA as a tool for learning with particular focus on how to frame their learning process by using the theory of Scaffolding as an approach.

Over all aim

1) Analyse teachers' underlying factors of motivation for using PA as a learning tool using The Self Determination Theory (SDT), and 2) analyse how to support teachers' motivation by using the theory of scaffolding.

This objective will be investigated through the following research questions:

* What type of motivation structures and patterns from The Self-Determination Theory occur when using PA as a tool for learning?
* How and why are elements such as didactics, the learning environment and professional identification important and furthermore how do they relate to teachers' motivation?
* How can motivation be supported and framed by using the theory of scaffolding?

The goal is to: 1) Reach a systematic view and understanding of motivation by analysing how it affects teachers' use of PA as a tool for learning; 2) understand how to maintain and support motivation; 3) offer new and scientifically based knowledge for working with PA in a school context particularly for teachers responsible for developing and engaging in PA; and 4) offer teachers an insight into their own motivation towards PA.

Self-Determination Theory As a tool for analysing the patterns and structures of motivation The Self-Determination Theory (SDT) is used. The SDT is highly suitable when analysing underlying factors of motivation within an individual, and will be used as a starting point for understanding the elements of the teachers' motivation - both intrinsically and extrinsically.

According to Deci and Ryan, who developed the model, all human motivation is based on three innate psychological needs: competence, autonomy and relatedness. In this theory the distinction between self-determined or autonomous and controlled types of motivation will offer a way of measuring structures and patterns related to the teachers motivation focusing on motivation as an psychological process. These different types of motivation (autonomous and controlled) reflect individual reasons for participating in activities: autonomous is defined as engaging in an activity because it is perceived to be consistent with intrinsic goals. In contrast, controlled means engaging in an activity for external reasons such as rewards or approval from others. The model offers four types of extrinsic motivation: external, introjected, identified and integrated. These four types of extrinsic motivation are viewed as a motivation process from external to internal regulation. Using these four types of extrinsic motivation, it is possible to understand what kind of motivation patterns and structures occur when using PA and furthermore enable a nuanced look at teachers' intrinsic or extrinsic motivation for using PA as a tool for learning.

Scaffolding motivation- and learning processes By using elements from the scaffolding theory, it is examined how to support and maintain motivation in a learning process where PA is implemented. The method was originally developed as a way of examining children's learning processes, however, in previous research on this area, it was found that scaffolding teachers is equally important as scaffolding children in a learning process - especially when the learning process is new. The approach or method of scaffolding is basically a way of framing and supporting a learning process dividing it into six levels. Wood, Bruner and Ross pointed out that all learning processes require some sort of scaffolding where a more competent person offers support in the learning process using the appropriate amount of structure and guidance. By using this method, it is possible to point out how and where to support teachers in the process of developing and integrating PA and furthermore to point out, based on the findings from the SDT, how to support and more importantly to maintain teachers motivation for using PA as a tool for learning. In this sense the teacher is viewed as the learner undergoing a learning process. Inspired by the Russian psychologist Lev Vygotski's theory of The Zone of Proximal Development, Wood, Bruner & Ross identified six levels of scaffolding. The six levels are: 1) Recruitment - gaining the interest from the learner; 2) Reduction in the degrees of freedom - simplifying the task; 3) Direction maintenance - keeping the learner on track; 4) Marking of critical features - marking the relevant and irrelevant parts of the task; 5) Frustration control - offering support and guidance; and 6) Demonstration - showing the learner the solution.

Research design The research design in this Ph.D. project uses mixed methods and is based on the methods mentioned below. Applying these different types of both quantitative and qualitative methods, it is possible to examine and analyse the objectives from different angles making sure that the point of data saturation is reached and at the same time answer the over all aim and research questions. This Ph.D. project does not contain a comparative study, but instead focus on gaining a deep insight into what is at stake regarding teachers' motivation after the implementation of the Danish School Reform.

1. A thorough literature review based on current national and international literature will be carried out. This will be conducted in accordance to the key research questions of this project.
2. Survey: A survey will provide a basic knowledge of teachers' motivation and furthermore give the opportunity to define teachers' motivation based on the SDT. The questionnaire will be distributed to minimum 500 teachers in Denmark, who will be selected from a variety of Danish Public Schools based on the following criteria: Size, location, and socio-demographics.

   The sample will consist of key respondents (teachers) that potentially will provide the data that will make it possible to answer the main objectives of this Ph.D. project and at the same time make sure that maximum variation is obtained. Teachers will therefore be selected based on the following differentiation, where teachers from both categories are needed: Age, gender, subject, class and experience.

   The questionnaire will be based on the The Work Task Motivation Scale for Teachers (WTMST).
3. Based on the knowledge gained from the questionnaires, where it is defined how the selected teachers are motivated in-depth interviews will be conducted with 10 teachers. The sample will consist of teachers that show different levels of both intrinsic and extrinsic motivation in accordance to the SDT and picked from the survey.

ELIGIBILITY:
Inclusion Criteria:

* teachers across age, gender, subject, class and experience

Exclusion Criteria:

* members of school management, students

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Danish school teachers in the public school system
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
teachers' motivation based on the Self-Determination Theory | January 2017 - June 2017
  Survey instrument based on the Self-Determination Theory

SECONDARY OUTCOMES:
teachers' need for scaffolding | August 2017 - december 2017
  Personal interviews with selected teachers.

CONTACTS AND LOCATIONS:
Overall Officials: Jørgen Povlsen, Study Director — University of Southern Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Knudsen LS, Skovgaard T, Bredahl T. Understanding and scaffolding Danish schoolteachers' motivation for using classroom-based physical activity: study protocol for a mixed methods study. BMJ Open. 2018 Mar 14;8(3):e019857. doi: 10.1136/bmjopen-2017-019857. PMID 29540419
- See also: Louise Stjerne Knudsen - profile — http://findresearcher.sdu.dk/portal/en/persons/louise-stjerne-knudsen(82021dca-c7e0-4f60-8f0e-da84ddc9ee77).html